CLINICAL TRIAL: NCT05365776
Title: Graded Exposure Therapy for Fear Avoidance Behaviour (GET FAB) After Concussion
Brief Title: Graded Exposure Therapy for Fear Avoidance Behaviour After Concussion
Acronym: GET-FAB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H21-02605
Record Dates: First submitted 2022-03-10; First posted 2022-05-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the study hypotheses and treatment arms, but not to the type of intervention they are receiving. Outcome assessors will be blinded to participants' treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Graded Exposure Therapy (Experimental)
  Interventions: Behavioral: Graded Exposure Therapy
- Arm 2: Prescribed Aerobic Exercise (Active Comparator)
  Interventions: Behavioral: Prescribed aerobic exercise
- Arm 3: Enhanced usual care (Active Comparator)
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: Graded Exposure Therapy — Graded exposure therapy is delivered by a psychologist over 12 individual (1:1) secure videoconference sessions. The core active ingredient is graded situational exposure to foster habituation and challenge beliefs that the avoided activities are dangerous. Homework exercises involve planned exposure exercises in the home and community to support generalization.
  Arms: Arm 1: Graded Exposure Therapy
Behavioral: Prescribed aerobic exercise — Participants will be asked to complete 30 minutes of aerobic exercise on 5 days/week for a 12-week period. Participants select the mode (e.g., swimming, jogging, bicycling) and location of exercise (e.g., outdoors, a gym or community centre, at home). The initial exercise intensity target will be based on the Buffalo Concussion Bike Test. The target progression will be 3-5 beats per minute every two weeks.
  Arms: Arm 2: Prescribed Aerobic Exercise
Other: Enhanced usual care — Usual care (education about concussion from the website: concussion.vch.ca/) will be enhanced through email message support.
  Arms: Arm 3: Enhanced usual care

SUMMARY:
Concussions are very common. Although many people recover well from concussion, some will have persistent symptoms and difficulties with daily activities. How people cope with their symptoms following concussion powerfully influences their recovery. Fear avoidance behaviour is a particularly unhelpful approach to coping, in which people perceive their pre-injury activities as unnecessarily dangerous and take great care to avoid overexertion and overstimulation. The investigators developed and pilot tested a behavioural therapy, called graded exposure therapy, to reduce fear avoidance behaviour. Our preliminary work suggested that graded exposure therapy was acceptable to patients with concussion and possibly beneficial for their recovery. The GET FAB after concussion study will assess the effectiveness of graded exposure therapy.

DETAILED DESCRIPTION:
GET FAB is a multisite randomized controlled trial designed to evaluate a behavioural treatment (graded exposure therapy) for adults with persistent symptoms after concussion. Participants in this study will be recruited from a network of concussion clinics in Canada. This study follows from the investigators' prior work establishing that (1) fear avoidance behaviour is a risk factor for poor concussion outcome, (2) graded exposure therapy reduces fear avoidance behaviour, and (3) graded exposure therapy is perceived as credible and is well-tolerated by patients with persistent post-concussion symptoms.

Participants will be assigned at random (in a 1:2:2 ratio) to receive enhanced usual care, graded exposure therapy group, or another therapy that might have similar benefits (prescribed aerobic exercise). The investigators hypothesize that patients who participate in graded exposure therapy will have reduced fear avoidance behaviour and improved daily functioning compared to other treatment conditions and this difference will be greatest for patients who enter the study with high fear avoidance behaviour.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-70 years;
2. sustained a concussion according to the ACRM mTBI Task Force definition between 1 and 24 months ago
3. fluent in English, because validated translations are not available for most questionnaires and recruiting multilingual therapists is not feasible;
4. access to a computer, tablet, or smartphone with internet capability;
5. 3 or more moderate-severe symptoms on the Rivermead Postconcussion Symptom Questionnaire.

Exclusion Criteria:

1. medical contraindication to aerobic exercise (cardiac disease, chest pain with exertion, acute bone/joint/soft tissue injury aggravated by exercise)
2. change in cardiac medication within the last month, such as beta blockers, calcium channel blockers, or ivabradine
3. involved in personal injury litigation for index mTBI
4. currently pregnant or plan to become pregnant within the next three months
5. severe/unstable medical or psychiatric condition that could worsen over the next year")

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post Concussion Symptoms Questionnaire (RPQ): Change | 3 months
  Score of 0-64, with a higher score indicates worse symptoms.

SECONDARY OUTCOMES:
Fear Avoidance Behaviour after Traumatic Brain Injury Questionnaire (FAB-TBI): Change | 3 months
  score of 0-48, where higher score indicates higher avoidance.

OTHER OUTCOMES:
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 12-item: interviewer version: Change. | 3 months
  score of 12 to 60, where higher scores indicate higher disability or loss of function
The Generalized Anxiety Disorder-7 | 3 months
  score of 0-15, where higher scores indicate severity of anxiety experienced.
Personal Health Questionnaire-9 | 3 months
  score of 0-27, where higher scores indicate severity of depression experienced.
The Post-Concussion Functional Scale-Screen | baseline and 3 months
  0 (unable) - 5 (more than 2 hours), higher score means longer length of time an activity can be tolerated without symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (7):
- Canada (7):
  - Calgary Brain Injury Program, Calgary, Alberta
  - Fraser Health Acquired Brain Injury and Concussion Services, Langley, British Columbia
  - G.F. Strong Adult Concussion Services, Vancouver, British Columbia
  - Sunnybrooke Traumatic Brain Injury Clinic, Toronto, Ontario
  - Head Injury Clinic at St. Michael's, Toronto, Ontario
  - Hull-Ellis Concussion and Research Clinic, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data (including data dictionaries).
Time Frame: Immediately following publication. No end date.
Access Criteria: Upon reasonable request. Requests can be made to the Principal Investigator.

REFERENCES:
- [Background] Silverberg ND, Cairncross M, Brasher PMA, Vranceanu AM, Snell DL, Yeates KO, Panenka WJ, Iverson GL, Debert CT, Bayley MT, Hunt C, Baker A, Burke MJ; Canadian Traumatic Brain Injury Research Consortium (CTRC). Feasibility of Concussion Rehabilitation Approaches Tailored to Psychological Coping Styles: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1565-1573.e2. doi: 10.1016/j.apmr.2021.12.005. Epub 2021 Dec 28. PMID 34971596
- [Derived] Mikolic A, Klotz T, Brasher P, Yeates K, Vranceanu AM, Kendall KD, Snell DL, Debert CT, Bayley M, Panenka W, Cairncross M, Hunt C, Burke M, Tartaglia MC, Silverberg N; Canadian Traumatic Brain Injury Research Consortium (CTRC). Graded Exposure Therapy for Fear Avoidance Behaviour After Concussion (GET FAB): protocol for a multisite Canadian randomised controlled trial. BMJ Open. 2024 Jul 1;14(6):e086602. doi: 10.1136/bmjopen-2024-086602. PMID 38950993